CLINICAL TRIAL: NCT05314803
Title: Yoga for Young Adults Affected by Cancer: Exploring Implementation and Effectiveness of an Online Program
Brief Title: Yoga for Young Adults Affected by Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-20-0098 (sub-study)
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-02

CONDITIONS: Young Adult Cancer; Young Adult Oncology
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga (Experimental): Participants receive online, group-based yoga classes 2 times/week for 60 minutes/class over 12 weeks.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Participants receive the yoga program, which is delivered by a trained yoga instructor (completed at least a 200-hour yoga teacher training, Yoga Thrive Teacher Training Certification (or similar), and/or practical experience working with individuals affected by cancer). The first class of the week is comprised of 45 minutes of gentle, progressive, hatha-based yoga sequencing and postures with the last 15 minutes focused on guided behaviour change and mindfulness techniques that varies week-to-week, based on the participants in the class. The second class of the week is 60 minutes of gentle, yin-based yoga sequencing and postures with an element of opening and relaxing.

SUMMARY:
Yoga may enhance physical and psychological outcomes among young adults affected by cancer. Yet, yoga has rarely been studied in this population. We developed and piloted a yoga program, which is now ready for implementation and evaluation. This single-group, mixed-methods project will explore effectiveness and implementation of the yoga program.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 years or older;
2. Diagnosed with cancer between the ages of 18-39 years;
3. At any stage of their cancer experience (i.e., on- or off-treatment);
4. Able to safely engage in yoga, as assessed by completing the Get Active Questionnaire and obtaining medical clearance (if indicated).
5. Willing and able to complete informed consent, questionnaires, physical assessments, and an interview in English.

Exclusion Criteria:

1. Previous enrolment in the study, to avoid contamination and/or ceiling effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Reach | Through study completion, an average of 5 years
  The number of people who participate, and reasons why or why not.

SECONDARY OUTCOMES:
Attendance | Through study completion, an average of 5 years
  Number of classes attended out of the number of classes offered by study staff.
Adherence | Through study completion, an average of 5 years
  Number of classes attended out of the number of classes offered by study staff.
Missing data | Through study completion, an average of 5 years
  Percentage of missing data on quantitative measures and completion of qualitative interviews.
Barriers and facilitators to exercise participation | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in Barrier Self-Efficacy Scale (1). Scale range 0-100; higher scores indicates less barriers to participation.
Physical activity levels | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Changes in Godin Leisure Time Scale (2). Individuals indicate how many times per week and how long per session they exercise at certain intensity (mild, moderate, high). Higher scores indicate higher levels of physical activity.
Fatigue | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (3). Scale range 0-4; selected items are reverse scored; higher score indicate less fatigue.
Cognition | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Changes in Functional Assessment of Cancer Therapy - Cognitive Scale (4). Scale range 1-4; some items are reversed scored; higher scores indicate less cognitive impairment.
Cancer-related symptoms | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in Edmonton Symptom Assessment Scale (5). Scale range 0-10; lower scores indicate fewer/less severe symptoms.
General health-related quality of life | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in EuroQual - 5Dimensions (EQ-5D) Scale (6). Scale range 1-5 with lower scores indicating greater quality of life; visual analogue scale range 0-100 with higher scores indicating greater quality of life.
General well-being | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in Functional Assessment of Cancer Therapy - General Scale (7). Scale range 0-4; selected items are reversed scored; higher scores indicate greater quality of life.
Mindfulness | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in Mindful Attention Awareness Scale (8). Scale range 1-6; higher scores indicate higher levels of dispositional mindfulness.
Self-compassion | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in Self-Compassion Scale (9). Scale range 1-5; higher scores indicate greater self-compassion.
Stress | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in Perceived Stress Scale (10). Scale range 0-4; some items are reverse scored; higher scores indicate more perceived stress.
Group identification | Post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in Group Identification Scale (11). Scale range 1-7; higher scores indicate greater identification with the group.
Balance | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in one legged stance test (seconds) (see 12).
Shoulder range of motion | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in active shoulder flexion range of motion (degrees) (see 12).
Lower extremity flexibility | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in sit-and-reach test (cm) (see 12).
Functional performance | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in sit-to-stand (number of repetitions in 30 seconds) (see 12).
Aerobic endurance | Baseline (week 0), post-program (week 12), 6-month follow-up (week 24), 1 year follow-up (week 52)
  Change in 2 minute step test (steps) results (see 12).
Adverse events | Through study completion, an average of 5 years
  Adverse events will be defined as any negative effect caused (or suspected to be caused by) the yoga program.
Time to implement and deliver | Through study completion, an average of 5 years
  Time and expertise to deliver the intervention and physical assessments will be tracked.
Yoga program fidelity | Through study completion, an average of 5 years
  Fidelity of the physical activity program implementation will be assessed via randomly video-auditing a subset of classes.

CONTACTS AND LOCATIONS:
Overall Officials: S. Nicole Culos-Reed, PhD, Study Director — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Rogers LQ, Courneya KS, Verhulst S, Markwell S, Lanzotti V, Shah P. Exercise barrier and task self-efficacy in breast cancer patients during treatment. Support Care Cancer. 2006 Jan;14(1):84-90. doi: 10.1007/s00520-005-0851-2. Epub 2005 Jul 9. PMID 16007455
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Acaster S, Dickerhoof R, DeBusk K, Bernard K, Strauss W, Allen LF. Qualitative and quantitative validation of the FACIT-fatigue scale in iron deficiency anemia. Health Qual Life Outcomes. 2015 May 17;13:60. doi: 10.1186/s12955-015-0257-x. PMID 25980742
- [Background] Wagner L, Sweet J, Butt Z, Lai J-S, Cella D. Measuring patient self-reported cognitive function: development of the functional assessment of cancer therapy-cognitive function instrument. J Support Oncol, 2009. 7(6): W32-W39.
- [Background] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Background] Pickard AS, De Leon MC, Kohlmann T, Cella D, Rosenbloom S. Psychometric comparison of the standard EQ-5D to a 5 level version in cancer patients. Med Care. 2007 Mar;45(3):259-63. doi: 10.1097/01.mlr.0000254515.63841.81. PMID 17304084
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Neff KD. Development and validation of a scale to measure self-compassion. Self Ident, 2003. 2: 223-50.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Sani F, Madhok V, Norbury M, Dugard P, Wakefield JR. Greater number of group identifications is associated with lower odds of being depressed: evidence from a Scottish community sample. Soc Psychiatry Psychiatr Epidemiol. 2015 Sep;50(9):1389-97. doi: 10.1007/s00127-015-1076-4. Epub 2015 Jun 10. PMID 26058588
- [Background] McNeely ML, Sellar C, Williamson T, Shea-Budgell M, Joy AA, Lau HY, Easaw JC, Murtha AD, Vallance J, Courneya K, Mackey JR, Parliament M, Culos-Reed N. Community-based exercise for health promotion and secondary cancer prevention in Canada: protocol for a hybrid effectiveness-implementation study. BMJ Open. 2019 Sep 13;9(9):e029975. doi: 10.1136/bmjopen-2019-029975. PMID 31519676
- [Derived] Wurz A, McLaughlin E, Janzen A, Cripps H, Huang L, Molina H, Cowley L, Dreger J, Culos-Reed SN, Quinn K, Currey IMOL, Pacelli MH, Coombs M, Shamshad S. A Protocol for a Mixed Methods, Single-Arm, Hybrid Effectiveness-Implementation Trial Evaluating a 12-week Yoga Intervention Delivered by Videoconference for Young Adults Diagnosed With Cancer. Glob Adv Integr Med Health. 2024 Dec 22;13:27536130241305130. doi: 10.1177/27536130241305130. eCollection 2024 Jan-Dec. PMID 39717073